CLINICAL TRIAL: NCT06317935
Title: The Effect of Virtual Reality Intervention on Upper Extremity Functioning and Perceived Independence in Daily Life in Children With Hemiplegic Cerebral Palsy
Brief Title: The Effect of Virtual Reality Application on Independence and Hand Functions in Daily Life in Children With CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Basak Karadag, Occupational Therapist, PhD Student, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: HU-ERG-BK-01
Record Dates: First submitted 2024-02-20; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Virtual Reality; Upper Extremity; Hemiplegic Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Two groups, intervention (A) and control (B), will be created from the target research group using the randomization method.
  Intervention group (A) will receive virtual reality application for 30 minutes, 5 days a week for 3 weeks, in addition to traditional occupational therapy and physiotherapy approaches for the first 3 weeks, and will receive only traditional treatments between 3-6 weeks.
  The control group (B) will receive only traditional occupational therapy and physiotherapy approaches for the first 3 weeks, and between 3-6 weeks, they will receive virtual reality application in addition to traditional approaches for 30 minutes, 5 days a week for 3 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ArmeoSenso (Other): ArmeoSenso virtual reality application will be applied to group A in the 0-3 weeks of the study and to group B in the 3-6 weeks.
  Interventions: Other: ArmeoSenso; Other: Traditional Rehabilitation
- Traditional rehabilitation (Other): Traditional rehabilitation (physiotherapy and occupational therapy) approaches will continue to be applied to groups A and B at all stages of the research.
  Interventions: Other: Traditional Rehabilitation

INTERVENTIONS:
Other: ArmeoSenso — ArmeoSenso is an upper extremity virtual reality application with three motion sensors and one hand grip sensor. The device detects the person's body, arm, forearm and hand movements and displays the reflection of the movements on the screen. The application includes studies on upper extremity functions.
  Arms: ArmeoSenso
Other: Traditional Rehabilitation — It includes traditional occupational therapy and physiotherapy approaches.

SUMMARY:
The aim of this study is to evaluate the effect of virtual reality applications on the level of independence and upper extremity functionality perceived by children in daily life in children with hemipegic cerebral palsy.

The research is a randomized controlled, cross-over study. The sample group of the research is children diagnosed with hemiplegic cerebral palsy and families who are receiving inpatient treatment in the pediatric service of Ankara City Hospital Physical Therapy and Rehabilitation Hospital.

Two groups, intervention (A) and control (B), will be created from the target research group using the randomization method.

The upper extremity functionality of both research groups before the intervention will be evaluated with the 'Motor Activity Diary for Children' scale and the perceived independence level with the 'Children's Hand Use Experience' scale.

After the initial evaluation is completed, group A, represented as the intervention group, will receive ArmeoSenso virtual reality intervention in the upper extremity hand function laboratory for 3 weeks, 5 days a week, each session for 30 minutes, in addition to traditional occupational therapy and physiotherapy rehabilitation programs. Meanwhile, group B, represented as the control group, will continue the traditional occupational therapy and physiotherapy rehabilitation program. At the end of the third week of the intervention, tests measuring upper extremity functionality and perceived independence level will be repeated.

Measurement tools will be repeated at the beginning of the intervention, at the end of the 3rd week, and at the end of the intervention.

DETAILED DESCRIPTION:
The sample group of the research is children between the ages of 6-12, diagnosed with hemiplegic cerebral palsy, who are receiving inpatient treatment in the pediatric service of Ankara City Hospital Physical Therapy and Rehabilitation Hospital, and their families.

Statistical power analysis was performed to calculate the number of people required to be included in the study. Statistical power analysis was performed with G*Power v.3.1.9.7 software. In the analysis, the Type 1 error margin (α) was accepted as 5% and the desired statistical power (1-β) was accepted as 0.80. In order to carry out the analysis, randomized controlled studies in the literature on the subject that reported effect sizes were examined. Studies have found that in virtual reality-based interventions applied to children with cerebral palsy, strong to very strong effect sizes were reported between intervention and control groups in variables such as upper extremity functions and performance in daily living activities (4, 7-11). When calculations were made using the strong effect size (Cohen's d = 0.80) in the sample size analysis, it was determined that the smallest sample size that needed to be reached for both groups was 26. Therefore, a total of 52 people were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* - Having a diagnosis of hemiplegic SP
* Being between the ages of 6-12
* Not having any fixed contracture in the upper extremity
* According to the Modified Ashworth Scale, the upper extremity spasticity value is at the level of 1,1+,2 or 3
* Being at level I, II or III according to the Gross Motor Function Classification System (GMFCS)
* Being at level II or III according to the Manual Ability Classification System (MACS)
* Being at level I, II or III according to the Communication Function Classification System (CFCS)
* Being within the normal cognitive level according to the Modified Pediatrics Mini Mental Test score
* Being at level I, II or III according to the Eating and Drinking Ability Classification System (EDACS)
* Being at level I, II or III according to the Visual Function Classification System for Children with Cerabral Palsy (VFCS)
* Volunteering to participate in the study

Exclusion Criteria:

* Having botolinum toxin injection within the last 6 months
* Having undergone a surgical procedure within the last 1 year
* Fracture, trauma, etc. in the upper extremity. to live

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-04-23 (Estimated); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
The effect of virtual reality applications on perceived independence in daily life in hemiplegic CP. | At the end of the 6th week
  The independence levels perceived by children with hemiplegic CP in daily life will be evaluated with the Children's Hand Use Experience Questionnaire.
The effect of virtual reality applications on upper extremity functionality in daily life in children with hemiplegic CP. | At the end of the 6th week
  The impact on the upper extremity functionality of children with hemiplegic CP in daily life will be evaluated with the Pediatric Motor Activity Log-Revised test.

SECONDARY OUTCOMES:
Dosimetry of virtual reality applications | At the end of the 6th week
  As suggested in further research, examining the dosimetric properties of virtual reality applications such as frequency and duration and comparing them with other studies.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Karadağ, MSc, Principal Investigator — Ankara City Hospital Bilkent; Meral Huri, Professor, Study Director — Hacettepe University; Berke Aras, Ass.Prof., Principal Investigator — Ankara City Hospital Bilkent; Özge Tezen, MD, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Multiple Locations, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only the principal investigator can access information about individuals; other researchers will not be able to access this information due to blinding.

REFERENCES:
- [Background] Chen YP, Lee SY, Howard AM. Effect of virtual reality on upper extremity function in children with cerebral palsy: a meta-analysis. Pediatr Phys Ther. 2014 Fall;26(3):289-300. doi: 10.1097/PEP.0000000000000046. PMID 24819682
- [Background] Goyal C, Vardhan V, Naqvi W. Virtual Reality-Based Intervention for Enhancing Upper Extremity Function in Children With Hemiplegic Cerebral Palsy: A Literature Review. Cureus. 2022 Jan 28;14(1):e21693. doi: 10.7759/cureus.21693. eCollection 2022 Jan. PMID 35237486